CLINICAL TRIAL: NCT06460064
Title: A Single Center, Randomized, Double-blind, Placebo-controlled, First-in-human Phase 1 Study to Assess the Safety, Tolerability and Immunogenicity of the Adjuvanted Universal Influenza Vaccine "fH1/DSP-0546LP" After Intramuscular (IM) Administrations in Healthy Adults
Brief Title: First-in-human Study to Assess the Safety, Tolerability and Immunogenicity of the Adjuvanted Universal Influenza Vaccine fH1/DSP-0546LP
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R2411201; JP19pc0101043 (Other Grant/Funding Number: Japan Agency for Medical Research and Development); 2023-504378-39-00 (Registry Identifier: Clinical Trials Information System)
Record Dates: First submitted 2024-04-29; First posted 2024-06-14 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Influenza
Keywords: Influenza; universal; vaccine; adjuvant; TLR7
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, Investigator staff, assessors, clinical operations personnel, data analysts, and personnel at central laboratories will remain blinded to the identity of the treatment from the time of randomization until clinical database lock and study unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- combination of fH1 2 ug and DSP-0546LP 2.5 ug (Experimental): The study vaccine (fH1 2 ug and DSP-0546LP 2.5 ug) will be administered IM into the deltoid muscle of the non-dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: fH1 2 ug; Biological: DSP-0546LP 2.5 ug
- combination of fH1 8 ug and DSP-0546LP 2.5 ug (Experimental): The study vaccine (fH1 8 ug and DSP-0546LP 2.5 ug) will be administered IM into the deltoid muscle of the non-dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: fH1 8 ug; Biological: DSP-0546LP 2.5 ug
- combination of fH1 2 ug and DSP-0546LP 5 ug (Experimental): The study vaccine (fH1 2 ug and DSP-0546LP 5 ug) will be administered IM into the deltoid muscle of the non-dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: fH1 2 ug; Biological: DSP-0546LP 5 ug
- combination of fH1 8 ug and DSP-0546LP 5 ug (Experimental): The study vaccine (fH1 8 ug and DSP-0546LP 5 ug) will be administered IM into the deltoid muscle of the non-dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: fH1 8 ug; Biological: DSP-0546LP 5 ug
- combination of fH1 2 ug and DSP-0546LP 10 ug (Experimental): The study vaccine (fH1 2 ug and DSP-0546LP 10 ug) will be administered IM into the deltoid muscle of the non-dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: fH1 2 ug; Biological: DSP-0546LP 10 ug
- combination of fH1 8 ug and DSP-0546LP 10 ug (Experimental): The study vaccine (fH1 8 ug and DSP-0546LP 10 ug) will be administered IM into the deltoid muscle of the non- dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: fH1 8 ug; Biological: DSP-0546LP 10 ug
- fH1 2 ug (Experimental): The study vaccine (fH1 2 ug) will be administered IM into the deltoid muscle of the non- dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: fH1 2 ug
- fH1 8 ug (Experimental): The study vaccine (fH1 8 ug) will be administered IM into the deltoid muscle of the non-dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: fH1 8 ug
- DSP-0546LP 2.5 ug (Experimental): The study vaccine (DSP-0546LP 2.5 ug) will be administered IM into the deltoid muscle of the non-dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: DSP-0546LP 2.5 ug
- DSP-0546LP 5 ug (Experimental): The study vaccine (DSP-0546LP 5 ug) will be administered IM into the deltoid muscle of the non- dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: DSP-0546LP 5 ug
- DSP-0546LP 10 ug (Experimental): The study vaccine (DSP-0546LP 10 ug) will be administered IM into the deltoid muscle of the non- dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: DSP-0546LP 10 ug
- Placebo (Placebo Comparator): The study vaccine (placebo) will be administered IM into the deltoid muscle of the non- dominant upper arm whenever possible. Subjects will receive 2 administrations at 3-week intervals.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: fH1 2 ug — 2 administrations at 3-week intervals.
  Arms: combination of fH1 2 ug and DSP-0546LP 10 ug; combination of fH1 2 ug and DSP-0546LP 2.5 ug; combination of fH1 2 ug and DSP-0546LP 5 ug; fH1 2 ug
Biological: fH1 8 ug — 2 administrations at 3-week intervals.
  Arms: combination of fH1 8 ug and DSP-0546LP 10 ug; combination of fH1 8 ug and DSP-0546LP 2.5 ug; combination of fH1 8 ug and DSP-0546LP 5 ug; fH1 8 ug
Biological: DSP-0546LP 2.5 ug — 2 administrations at 3-week intervals.
  Arms: DSP-0546LP 2.5 ug; combination of fH1 2 ug and DSP-0546LP 2.5 ug; combination of fH1 8 ug and DSP-0546LP 2.5 ug
Biological: DSP-0546LP 5 ug — 2 administrations at 3-week intervals.
  Arms: DSP-0546LP 5 ug; combination of fH1 2 ug and DSP-0546LP 5 ug; combination of fH1 8 ug and DSP-0546LP 5 ug
Biological: DSP-0546LP 10 ug — 2 administrations at 3-week intervals.
  Arms: DSP-0546LP 10 ug; combination of fH1 2 ug and DSP-0546LP 10 ug; combination of fH1 8 ug and DSP-0546LP 10 ug
Biological: Placebo — 2 administrations at 3-week intervals.
  Arms: Placebo

SUMMARY:
This study is a single center, randomized, double-blind, placebo-controlled, dose-finding, FIH, Phase 1 study to assess the safety, tolerability, and immunogenicity of the adjuvanted Universal Influenza Vaccine (fH1/DSP-0546LP) after IM administrations in healthy adults.

DETAILED DESCRIPTION:
This will be a single center, randomized, placebo-controlled, double-blind study. In this study, safety, tolerability, and immunogenicity of fH1 formulated with DSP-0546LP will be assessed after IM administration in healthy adults aged 18 to 40 years.

This study includes 6 cohorts, with a combination of 2 dose levels of fH1 (2 and 8 μg), 3 dose levels of DSP-0546LP (2.5, 5, and 10 μg), and placebo. Each dose level of fH1 will be combined with the low, medium, and high dose level of DSP-0546LP. Subjects will receive 2 administrations at 3-week intervals.

Randomized subjects will undergo 11 visits including screening, 2 administration visits (Day 1 and Day 22 [± 2]), and follow-up visits on Day 4 (+1) (telephone contact), Day 8 (± 1), Day 25 (+1) (telephone contact), Day 29 (± 1), Day 36 (± 2), Day 50 (± 4), Day 204 (± 7), and Day 386 (± 10).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female subject between 18 and 40 years of age at the time of informed consent.
2. Subject who is fully informed of and understands the objectives, procedures, anticipated side effects of the vaccine and risks of the study and who voluntarily provides written consent to participate in the study.
3. Subject's body weight is equal to or more than 50 kg, and body mass index is at least 18 kg/m2 but no more than 30 kg/m2 at screening.
4. Subject willing and able to comply with the study requirements, including laboratory tests and reporting symptoms.
5. A male subject with a female partner of childbearing potential must agree to use adequate and reliable contraception (e.g., using condom or have had vasectomy with proven sterility for male and using contraceptive agents, diaphragm, intrauterine devices (IUDs), or bilateral tubal ligation for female partner) from informed consent until at least 30 days after last administration of the study vaccine.
6. A female subject is eligible for this study if she is neither pregnant nor breastfeeding and 1 of the following:

   1. Of non childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in greater than or equal to 1 year).
   2. Of childbearing potential but has been and agrees to continue practicing highly effective contraception from informed consent until at least 30 days after the last administration. Highly effective methods of contraception include 1 or more of the following:

      * a female subject who is abstinent or have a sexual relationship with sole female partner;
      * male partner who is sterile (vasectomized) prior to the female subject's entry into the study and is the sole sexual partner for the female subject;
      * hormonal (oral, intravaginal, transdermal, implantable or injectable), which is associated with inhibition of ovulation;
      * an intrauterine hormone-releasing system;
      * an intrauterine device with a documented failure rate of < 1%;
      * bilateral tubal occlusion.
7. A female subject who is premenopausal and of childbearing potential must have a negative urine pregnancy-test result at screening, on Days 1 and 22.
8. Subject must agree not to donate sperm or eggs from informed consent until at least 30 days after last administration of the study vaccine.

Exclusion Criteria:

1. Subject with a history of clinically significant cardiovascular, hepatic, renal, endocrine, gastrointestinal, hematological, respiratory, psychiatric or neurologic disease, and who is considered ineligible for the study by the Principal Investigator (PI) or sub Investigator.
2. Subject with other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior that may increase the risk of study participation or, in the Investigator's judgement, make the subject inappropriate for the study.
3. Subject immunocompromised with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
4. Subject with a history or evidence of autoimmune disease or known immunodeficiency of any cause or severe allergy.
5. Subject who receives chronic treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, e.g., for cancer or an autoimmune disease, within 60 days before the Screening Visit or planned receipt throughout the study. If systemic corticosteroids have been administered short term (< 14 days) for treatment of an acute illness, subjects should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before first administration. Inhaled/nebulized, intra articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
6. Subject with a history of severe adverse reaction associated with a vaccine and/or a known or suspected allergic reaction (e.g., anaphylaxis) or hypersensitivity to any component of the investigational product including egg protein.
7. Subject with a history of substance abuse or drug abuse. If there is any doubt about the correctness of the information provided by the subject (history) or observation of a behavior that raises concerns about drug use, drug screening will be conducted at the Screening Visit or prior to first administration.
8. Subject with a positive serology (hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus antigen/antibody) at screening.
9. Subject with any clinically significant abnormal clinical laboratory value (hematology, serum chemistry, urinalysis, coagulation) determined by the PI or sub-Investigator at screening.
10. Subject with a history of excessive alcohol consumption (defined as drinking at least 21 units of alcohol beverage per week for a man and 14 units of alcohol beverage per week for a woman) within 6 months of the Screening Visit. Following common drinks contain 1 unit of alcohol: 300 ml beer [4% alcohol by volume (ABV)], 100 ml of wine (12% ABV), 30 ml of spirits (40% ABV).
11. Subject who drinks large quantities of caffeinated beverages (coffee, tea, green tea, cola, tonic drink, etc) (approximately 1.8 L daily or more).
12. Subject with a history of tobacco (including electronic cigarette) dependency or subject who smokes ≥ 20 cigarettes daily (excluding subject who stopped smoking more than 2 years ago).
13. Subject who has received seasonal flu vaccine within a year prior to the Screening Visit.
14. Subject who has experienced significant blood loss or donated blood (≥ 400 mL) within 90 days prior to the first administration or donated 200 mL of blood or more within 30 days prior to the first administration; has donated blood components within 14 days prior to the first administration.
15. Subject who has received blood/plasma products or immunoglobulins within 6 months prior to the Screening Visit.
16. Subject who has received any investigational drug or who is currently participating or has participated in a clinical study within 90 days prior to the Screening Visit.
17. Subject who has participated in a clinical study of any influenza vaccine, or any investigational vaccine or experimental influenza viral challenge delivered directly to the respiratory tract within a year prior to the first administration.
18. Subject with a history of hospitalization (excluding hospitalization for medical checkup) for at least one night within 45 days prior to the Screening Visit.
19. Subject who has used prescription or over-the-counter medications except chronic medication and contraceptives for female subjects within 7 days or 5 half-lives prior to the first administration.
20. In the Investigator's judgement, the subject has current symptoms suggestive of an acute infection, or presence of long-term medical, neurologic, or psychiatric sequalae of prior COVID-19.
21. Subject who has received any other licensed vaccine within 28 days prior to screening or who is planning to receive any vaccine up to 28 days after the last vaccine administration.
22. Subject who is a staff member of the clinical site/Sponsor/Contract research organization (CRO) or the relative of a staff member.
23. Subject who is in the opinion of the PI or sub-Investigator, unsuitable in any other way to participate in this study.
24. Subject with bleeding disorder that would, in the opinion of the Investigator, contraindicate IM injection.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of solicited local adverse events (AEs) during a 7-day follow-up period after each administration. | 7 days after each administration
  Solicited local AEs: pain, redness, swelling, induration, warmth, and pruritus at injection site
Incidence of solicited systemic AEs during a 7-day follow-up period after each administration. | 7 days after each administration
  Solicited systemic AEs: feverishness, chills, myalgia, fatigue, headache, nausea, arthralgia, malaise, and body temperature (measured axillary)
Incidence of unsolicited AEs from the first administration to 4 weeks after the second administration. | From the first administration to 4 weeks after the second administration.
  Clinical observations, clinical laboratory values and vital signs
Incidence of serious adverse events (SAEs), AEs leading to study discontinuation, and adverse events of special interest throughout the study period. | From the first administration to 52-week follow-up after the second administration

SECONDARY OUTCOMES:
Percentage of subjects with increased immunoglobulin (Ig) G response to long alpha helix (LAH) after administration of fH1/DSP-0546LP. | From the day of the first administration to 52-week follow-up after the second administration
Percentage of subjects with increased neuraminidase inhibition antibody titer after administration of fH1/DSP-0546LP. | From the day of the first administration to 1 week after the second administration.
Seroconversion rate (SCR) of hemagglutination inhibition (HAI) antibody titers after administration of fH1/DSP-0546LP. | From the day of the first administration to 1 week after the second administration.
  SCR is defined as the percentage of subjects with either a baseline (Day 1) HAI titer < 1:10 and post-administration titer ≥ 1:40, or baseline titer ≥ 1:10 and ≥ 4-fold increase in post-administration titer.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Vaccinology, Ghent, Corneel Heymanslaan 10, Belgium